CLINICAL TRIAL: NCT03984981
Title: Brain Death Diagnosis at an Academic Tertiary Medical Care Center
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00244; me19Sutter4
Record Dates: First submitted 2019-05-06; First posted 2019-06-13 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Brain Death
Keywords: diagnosis of brain death
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of process required to diagnose brain death in adult patients — Assessment of process required to diagnose brain death in adult patients (demographics, clinical, laboratory, imaging, and treatment data). No questionnaires or study visits will be used.

SUMMARY:
The aim of this study is to assess and survey the quality of the process required to diagnose brain death in adult patients. This study of adult patients diagnosed brain dead or suspected of having brain death on the ICUs at the University Hospital Basel will be purely observational.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected and/or diagnosed brain death
* adults 18 years and over

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all adult (18 years or older) patients in whom brain death was suspected and/or diagnosed on the ICUs of the University Hospital Basel between January 1st 2008 and January 31st 2019.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
adherence to the local brain death protocol ( = measurement tool) for the process of brain death diagnosis | single time point assessment at baseline (after suspected brain death)
  the local brain death protocol ( = measurement tool) requires 1.) exclusion of the following conditions:
  * shock (mean arterial blood pressure > 60 mmHg, lactate < 4 mmol/l)
  * hypothermia (temperature > 35°C)
  * severe acidosis (pH > 7.3)
  * hyperosmolarity (osmolarity < 320 mmol/l)
  * severe electrolyte disorders (sodium > 125 mmol/l, phosphate > 0.3 mmol/l)
  * hypoglycemia (glucose > 4 mmol/l)
  * hyperammonemia (ammonia < 60 mumol/l)
  * uremia (urea < 25 mmol/l)
  * prolonged effects of medication (muscle relaxants, sedatives, recreational drugs)
  * severe hypothyreosis
    2.) clinical examination confirming:
  * fixed pupils (dilated or mid-dilated bilaterally)
  * absent vestibulo-ocular reflex
  * absent corneal reflex bilaterally
  * no reaction to painful stimulus bilaterally
  * absence of cough and gag reflex
  * absence of spontaneous breathing (apnea test)

SECONDARY OUTCOMES:
number of physicians involved | single time point assessment at baseline (after suspected brain death)
  number of physicians involved in the diagnostic procedures
frequency of ancillary tests performed | single time point assessment at baseline (after suspected brain death)
  frequency of ancillary tests (i.e. transcranial doppler ultrasound, computed tomography, magnetic resonance tomography, digital substraction angiography, electroencephalogram, somatosensory evoked potentials) performed
number of work-ups excluding suspected brain death | single time point assessment at baseline (after suspected brain death)
  number of work-ups excluding suspected brain death
number of diagnostic work-ups with insufficient performance and/or documentation | single time point assessment at baseline (after suspected brain death)
  number of diagnostic work-ups with insufficient performance and/or documentation
years of clinical experience of physicians involved | single time point assessment at baseline (after suspected brain death)
  years of clinical experience of physicians involved in the diagnostic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. med, Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (1):
- Clinic for Intensive Care Medicine, University Hospital Basel, Basel, Switzerland